CLINICAL TRIAL: NCT06807827
Title: Pharmacist-Led Educational Intervention for Diabetic Patients: a Randomized Interventional Trial to Evaluate the Impact on Medication Adherence and Quality of Life
Brief Title: Pharmacist-Led Cognitive Behavioral Intervention for Diabetic Patients: a Randomized Interventional Trial to Evaluate the Impact on Medication Adherence and Quality of Life
Acronym: COGNIPHARM-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Matti Ullah, Assistant Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MU0624-IF
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabete Mellitus
Keywords: Educational Intervention; Cognitive behavioral therapy; Pharmacist; Medication Adherence; Quality of life
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be entertained as part of their regular appointment for prescription filling without any information of which group they are assigned in. Moreover, following intervention, the outcomes will be assessed by the investigator who will be blinded about the participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Routine healthcare practices and protocols for diabetes management. Regular advice on medication, diet, and lifestyle modifications in accordance with established guidelines, Follows conventional approaches. Lifestyle Modification(Provide guidance on how to maintain a healthy lifestyle, including balanced diet, exercise and regular sleep patterns). General Knowledge advancement. General knowledge about disease and medicine. Pill planner will be provided to keep them adherent to their medication. General Medication counselling.
  Interventions: Other: Basic Education
- Cognitive Behavioral Interventional Group (Experimental): Specific Patient-centered strategies beyond routine care designed to address individualized needs. Customized interventions, including pharmacist-led educational sessions, personalized counseling, or advanced lifestyle modifications. Aims to enhance patient outcomes by providing tailored and innovative solutions for better diabetes management.
  Change in lifestyle / link with any daily activity (Yoga and Meditation Specifically guide about food portions and how to balance each food group in daily routine along with recommended daily physical activity type and duration. Pill planner will also be provided to this group.
  Medication counselling, Insulin technique, Dose Adjustment, Titration, Insulin Correction.
  Cognitive Behavioral Therapy will be provided.
  Interventions: Behavioral: Pharmacist-led Cognitive Behavioral therapy

INTERVENTIONS:
Behavioral: Pharmacist-led Cognitive Behavioral therapy — Pharmacist-led Cognitive Behavioral therapy is patient centered approach that focus both physical and emotional aspect of health is provided. It is focused to identify negative and change negative thought pattern and behavior to improve mental and physical well being.Incorporation education about healthy meal choices, relaxation techniques, self management strategies,to improve education about potential adverse effect, how to recognize and on followup calls how to adjust medication doses along with this is provided.
  Arms: Cognitive Behavioral Interventional Group
Other: Basic Education — Basic Education about lifestyle Modification(Provide guidance on how to maintain a healthy lifestyle, including balanced diet, exercise and regular sleep patterns). General Knowledge advancement. General knowledge about disease and medicine. Pill planner will be provided to keep them adherent to their medication. General Medication counselling.
  Arms: Control Group

SUMMARY:
This interventional study will to assess the impact of pharmacist-led educational intervention along with cognitive behavioral intervention in diabetic patients. Participants of this study will be provided regular counselling or cognitive behavioral intervention and educational material as part of their routine pharmacy visit. Researchers will compare the two groups to see which of the two groups improve in term of medication adherence and quality of life.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether incorporating pharmacist-led educational interventions along with Cognitive Behavioral Therapy (CBT) can result in better outcomes for diabetic patients. Effective diabetes management requires proper education and adherence to medication. Missed doses or irregular medication use can lead to poor glycemic control and increased complications. The study will examine if educational interventions along with Cognitive Behavioral Therapy (CBT) can have a favorable effect on various aspects of diabetes management coping techniques, Medication beliefs, reduction in hypo and hyperglycemic frequency, HbA1c and medication related problems (MRPs) medication adherence and overall quality of life of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

All confirmed Type II diabetic patients who visit endocrinology OPD Clinic during study duration.

Patients having HbA1c >8%. Follow up as well as new patients were included subjects willing to participate in the study with or without other severe co-morbidities were included in the study.

Exclusion Criteria:

GDM diabetic patients Patients with Central Obesity Type I DM Patients Patients with inadequate medical history Patient having HbA1c <8% Patient who are not interested in the study are excluded.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence score | 3 months
  Adherence will be assessed using (Medication Adherence Reporting Scale) MARS-10.
  This scale describes three-dimension, Medication adherence behavior (1-4), attitude towards taking medication (5-8), negative side effects and attitudes to psychotropic medication (9-10). Each question has Yes and No response, a response consistent with adherence is coded as 1 and with non-adherence coded as 0. Higher the score higher will be the adherence. Adherence <6 is poor adherence, and >8 is high adherence.
Quality of life Score | 3 months
  Patient's quality of life will be assessed using Revised Version of DQOL (RV-DQOL13 ; Audit of diabetes dependent quality of life) will be used to access the quality of life of the patient. Its scoring ranges from 1- 100

SECONDARY OUTCOMES:
Incidence of Drug-Drug Interactions | 3 months
  Drug interactions among oral anti glycemic and other drugs will be assessed using standard website (update-Lexicomp) It is used to access the reduction in no. of drug drug interaction after pharmacist intervention in both control and Cognitive Behavioral Intervention groups.
HbA1c % | 3 months
  HbA1c levels (%) will be assessed before the intervention is provided and after 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa International Hospital, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The sharing will be dependent on the consent provided by the patient.